CLINICAL TRIAL: NCT06237491
Title: Phase I, Open-Label Study of the Safety and Dosimetry of a 3-Dose Regimen of Escalating Doses of 177Lu-LNC1003 Injection in Adult Patients With Prostate Specific Membrane Antigen (PSMA)-Positive Metastatic Castration-Resistant Prostate Cancer (mCRPC)
Brief Title: The Safety and Dosimetry Study of 177Lu-LNC1003 Injection
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Yantai LNC Biotechnology Singapore PTE. LTD. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 177Lu-LNC1003-001
Record Dates: First submitted 2024-01-23; First posted 2024-02-01 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-03

CONDITIONS: Metastatic Castration-resistant Prostate Cancer, mCRPC

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Experimental: 177Lu-LNC1003 Injection group 1 (Experimental): 177Lu-LNC1003 Injection, a single dose of 30mCi will be administered every 6 weeks, for a total of 2 cycles.
  Interventions:
  Drug: 177Lu-LNC1003 Injection group 1 radionuclide therapy
  Interventions: Drug: 177Lu-LNC1003 Injection group 1
- Experimental: 177Lu-LNC1003 Injection group 2 (Experimental): 177Lu-LNC1003 Injection, a single dose of 50mCi will be administered every 6 weeks, for a total of 2 cycles.
  Interventions:
  Drug: 177Lu-LNC1003 Injection group 2 radionuclide therapy
  Interventions: Drug: 177Lu-LNC1003 Injection group 2
- Experimental: 177Lu-LNC1003 Injection group 3 (Experimental): 177Lu-LNC1003 Injection, a single dose of 70mCi will be administered every 6 weeks, for a total of 2 cycles.
  Interventions:
  Drug: 177Lu-LNC1003 Injection group 3 radionuclide therapy
  Interventions: Drug: 177Lu-LNC1003 Injection group 3

INTERVENTIONS:
Drug: 177Lu-LNC1003 Injection group 1 — The treatment regimen will consist of a single dose 30 mCi intravenous administration of 177Lu-LNC1004 Injection per 6-week cycle, for a total of 2 cycles, the dose per cycle will be fixed.
  Arms: Experimental: 177Lu-LNC1003 Injection group 1
Drug: 177Lu-LNC1003 Injection group 2 — The treatment regimen will consist of a single dose 50 mCi intravenous administration of 177Lu-LNC1004 Injection per 6-week cycle, for a total of 2 cycles, the dose per cycle will be fixed.
  Arms: Experimental: 177Lu-LNC1003 Injection group 2
Drug: 177Lu-LNC1003 Injection group 3 — The treatment regimen will consist of a single dose 70 mCi intravenous administration of 177Lu-LNC1004 Injection per 6-week cycle, for a total of 2 cycles, the dose per cycle will be fixed.
  Arms: Experimental: 177Lu-LNC1003 Injection group 3

SUMMARY:
This proposal is a phase I, open-label study of a 3-Dose Regimen of Escalating Doses of 177Lu-LNC1003 Injection in patients with PSMA-positive mCRPC.

In the clinical development, we aim to demonstrate the following:

1. Determination of the therapeutic dose(s) to be used in the expansion phase.
2. Demonstration of the safety and tolerability of 177Lu-LNC1003 at therapeutic doses.

The treatment regimen will consist of a single-dose intravenous administration of 177Lu-LNC1003 Injection per 6-week cycle, for a total of 2 cycles. The dose per cycle will be fixed for each patient and will be escalated in 3 different dose levels

DETAILED DESCRIPTION:
This proposal is a phase I, open-label study of a 3-Dose Regimen of Escalating Doses of 177Lu-LNC1003 Injection in patients with PSMA-positive mCRPC. The treatment regimen will consist of a single-dose intravenous administration of 177Lu-LNC1003 Injection per 6-week cycle, for a total of 2 cycles. The dose per cycle will be fixed for each patient and will be escalated in 3 different dose levels, from 30 mCi to 70 mCi (1.11 GBq - 2.59 GBq).

This classic "3+3" design recruits 3 patients for the first dose level group. If no dose limiting toxicity (DLT) occurs in the first cycle, then 3 new patients will enter the next higher dose level. If any DLT occurs at a certain dose level, 3 additional patients will be enrolled at this current dose level (in total 6 patients now) to be assessed. The highest dose level(s) at which less than one-third of patients (e.g., 0 of 3 or 1 of 6 patients) experience a DLT will be declared the maximum tolerated dose (MTD). If there is no MTD observed after the dose escalation up to 70 mCi, a comprehensive evaluation should be made by investigator and sponsor to determine whether an escalation to a higher dose can be conducted or not based on the known safety data, radiation doses for similar drugs documented in literature and treatment responses at the doses administered.

ELIGIBILITY:
Inclusion Criteria:

* Patients or authorized guardians must have the ability to understand and sign an approved informed consent form (ICF).
* Patients must have the ability to understand and comply with all protocol requirements.
* Patients must be aged 21 years or older.
* Patients must have histological, pathological, and/or cytological confirmation of PC that is refractory to or has progressed following prior treatments.
* Patients must have ≥ 1 metastatic lesion present on baseline and documented progressive mCRPC based on the Prostate Cancer Working Group 3 (PCWG3) criteria; patients must fill at least one of the following criteria:

  * PSA progression
  * Objective radiographic progression in soft tissue
  * New bone lesions
* Patients must have a castrate level of serum/plasma testosterone (< 50 ng/dL or < 1.7 nmol/L).
* Patients must have received treatment with at least one prior novel androgen receptor pathway inhibitor (such as enzalutamide, apalutamide, and/or abiraterone).
* Patients must have been deemed not suitable for chemotherapy, i.e., the patient refused chemotherapy or was judged unsuitable for chemotherapy by the doctor. Alternatively, patients may have been previously treated with at least one, but no more than two previous taxane regimens, or have been offered, but declined, or been ineligible for taxane-based chemotherapy. A taxane regimen is defined as a minimum exposure of 2 cycles of a taxane. If a patient has received only one taxane regimen, the patient is eligible if:

  a. The patient's physician deems him unsuitable to receive a second taxane regimen (e.g., frailty assessed by geriatric or health status evaluation, intolerance, etc.).
* Patients must have at least 1 measurable lesion as defined by Response Criteria in Solid Tumors (RECIST) version 1.1.
* Patients must be 68Ga-PSMA-11 PET/CT scan positive.
* Patients must have an Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1.
* Patients must have an adequate organ function, in the absence of clinical intervention within 28 days before the administration of the 177Lu-LNC1003, as defined by:

Hemoglobin (Hb) > 9.0g/dL White blood cell (WBC) count ≥ 3 x 109/L or absolute neutrophil count (ANC) >1.5 x 109/L Platelets ≥ 100 x 109/L International normalized ratio (INR) <1.5 for patients that are not on warfarin Prothrombin time (PTT) < 2 x ULN Total bilirubin <1.5 x ULN Serum albumin >3.0 g/dL Alanine aminotransferase (ALT) <3 x ULN, or<5 x ULN if deemed related to liver metastases from solid tumor Aspartate aminotransferase (AST) <3 x ULN, or<5 x ULN if deemed related to liver metastases from solid tumor Creatinine clearance ≥ 60 mL/min (calculated using the Cockcroft-Gault formula).

* All other toxicity parameters, except for alopecia, must be NCI-CTCAE v.5.0 Grade 0 or 1.
* Sexually active participants with female partners of childbearing potential are eligible to participate if they agree to follow 1 of the following methods of contraception consistently, starting from screening, during the study and for at least 14 weeks after the last dose of 177Lu-LNC1003 Injection:

Are abstinent from penile-vaginal intercourse as their usual and preferred lifestyle (abstinent on a long-term and persistent basis) and agree to remain abstinent; Are sterilized (with the appropriate post-vasectomy documentation of the absence of sperm in the ejaculate); Agree to use a male condom and have their partner use a contraceptive method with a failure rate of < 1% per year as described below when having penile-vaginal intercourse with a woman of childbearing potential who is not currently pregnant, and who agrees to the use of a condom by her partner.

* Participants must agree to refrain from donating sperm starting from Screening, during the study and for at least 14 weeks after the last dose of 177Lu-LNC1003 Injection.
* Sexually active participants with a pregnant or breastfeeding partner must agree to remain abstinent from penile vaginal intercourse; or use a male condom during each episode of penile penetration during the study.

Exclusion Criteria:

* Other identified malignancies within 5 years in addition to radically treated locally curable malignant tumors, such as basal or squamous cell skin cancer, superficial bladder cancer.
* Previous treatment with any of the following within 6 months before enrollment: Strontium-89, Samarium-153, Rhenium-186, Rhenium-188, Radium-223, hemi-body irradiation, 177Lu-PSMA-617 (Pluvicto) and any investigational beta-emitting radiotherapeutics.
* Any systemic anti-cancer therapy (e.g. PSMA-targeted radioligand therapy, chemotherapy, immunotherapy or biological therapy [including monoclonal antibodies]) within 28 days prior to day of enrollment
* Any investigational agents within 28 days of enrollment
* Other concurrent cytotoxic chemotherapy, immunotherapy, radioligand therapy, or investigational therapy
* Transfusion for the sole purpose of making a subject eligible for study inclusion
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to 177Lu-LNC1003 as assessed from medical records
* Participants who have not fully recovered from major surgery or significant traumatic injury prior to the first dose of study drug or expects to have major surgery during the study period or within 3 months after the last dose of study drug
* Life expectancy < 6 months as assessed by the treating physician
* Other serious illness(es) involving the cardiac, respiratory, CNS, renal, hepatic or hematological organ systems which might preclude completion of this study or interfere with determination of causality of any adverse effects experienced in this study
* A superscan; i.e., very high ratio of bone to background uptake due to high osteoblastic activity, as seen in the baseline Tc-99m diphosphonate bone scan.
* Clinically significant abnormalities on electrocardiogram (ECG) at screening including QTcF > 470 ms, and subjects who cannot tolerate high volume load.
* Active and clinically significant bacterial, fungal, or viral infections, including hepatitis B (HBV), hepatitis C (HCV), know human immunodeficiency virus (HIV), or acquired immunodeficiency syndrome (AIDS)-related illness (patients with treated HIV and hepatitis B or C could be included)
* Known brain metastases and/or carcinomatous meningitis, unless these metastases have been treated and stabilized
* Uncontrolled diabetes mellitus as defined by a HbA1c > 9%
* Prior external beam radiation therapy involving > 25% of the bone marrow
* Unmanageable urinary incontinence including physical outflow obstructions rendering the administration of 177Lu-LNC1003 unsafe.
* Unable to comply with relevant contact precautions post 177Lu-LNC1003 treatment.
* Any other condition, assessed by the investigator, that may increase the risk associated with study participation, interfere with the study interpretation, or in any other way make the subject unsuitable for participation in the study.

Min Age: 21 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-07 (Estimated); Primary Completion 2025-11-07 (Estimated); Study Completion 2025-12-17 (Estimated)

PRIMARY OUTCOMES:
the safety of 177Lu-LNC1003 Injection | through study completion, assessed up to 2 years.
  To evaluate the safety of 177Lu-LNC1003 Injection assessed from the number of patients with treatment-related adverse events using CTCAE v5.0.
To identify the dose-limiting toxicities (DLTs) | through cycle 1, an average of 6 weeks
  To identify DLTs of escalating doses of 177Lu-LNC1003 Injection up to 70 mCi (2.59 GBq) administered intravenously to patients in their first cycle of 6 weeks.
To determine if the MTD is among the explored dose levels and identify the expansion phase dose | Through study completion, assessed up to 2 years
  To determine if the maximum tolerated dose is among the explored dose levels and identify the recommended expansion phase dose of 177Lu-LNC1003 Injection.

IPD SHARING:
Plan to Share IPD: No